CLINICAL TRIAL: NCT05514236
Title: Effect of Virtual Reality and Music Therapy on Pain Relief in Outpatient Hysteroscopy: A Randomized Controlled Trial
Brief Title: Effect of Virtual Reality and Music Therapy on Pain Relief in Outpatient Hysteroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, YIP Ka Man, Principal Investigator, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRE 2022.237
Record Dates: First submitted 2022-08-16; First posted 2022-08-24 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Pain Management; Hysteroscopy
Keywords: Pain relief; Hysteroscopy
MeSH Terms: conditions — Agnosia | interventions — Virtual Reality Exposure Therapy; Music Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Virtual reality group (Experimental): Participants assigned to the Visual reality group will be given the virtual reality device (a headset) with immersive video content for use during the hysteroscopy. Designated moving objects with sound will be broadcasted on the screen to the participant in this group.
  Participant can adjust the volume of the sound according to her comfort.
  Interventions: Other: Virtual Reality Therapy
- Music group (Experimental): Participants in the music group will be given a headphone playing either classical light music or 'POP' songs according to their option during the hysteroscopy.
  Participant can adjust the volume of the sound according to her comfort.
  Interventions: Other: Music Therapy
- Control group (No Intervention): While participants in the control group will not be given any Virtual reality or music device.

INTERVENTIONS:
Other: Virtual Reality Therapy — Participants will be given the virtual reality device (a headset) with immersive video content for use during the hysteroscopy. Designated moving objects with sound will be broadcasted on the screen to the participant in this group.
  Participant can adjust the volume of the sound according to her comfort.
  Arms: Virtual reality group
Other: Music Therapy — Participants will be given a headphone playing either classical light music or 'POP' songs according to their option during the hysteroscopy.
  Participant can adjust the volume of the music according to her comfort.
  Arms: Music group

SUMMARY:
Outpatient hysteroscopy is an essential diagnostic procedure for abnormal uterine bleeding, such as menorrhagia or postmenopausal bleeding, to evaluate any intrauterine pathologies. It also serves as a therapeutic procedure such as removal of fibroids, polyps or intrauterine devices.However, the most common reason for procedure failure is pain.

On such occasions, the procedure has to be re-arranged in the operation theatre under regional or general anesthesia. Therefore, improvement in pain management can reduce patients' health care experience, patients' anesthetic and procedural risks, decrease healthcare costs, and reduce inconvenience to patients.

This randomized controlled trial aims at evaluating the effectiveness of non-pharmacological interventions (virtual reality and music therapy) in pain management during hysteroscopy. It can hopefully provide more clinical data to explore the role of non-pharmacological techniques in outpatient hysteroscopy pain control, hence help improve our participants' experience in outpatient hysteroscopy.

DETAILED DESCRIPTION:
Introduction:

Outpatient hysteroscopy is an essential diagnostic procedure for abnormal uterine bleeding, such as menorrhagia or postmenopausal bleeding, to evaluate any intrauterine pathologies. It also serves as a therapeutic procedure such as myomectomy, polypectomy and removal of lost intrauterine devices. However, the most common reason for procedure failure is pain. The frequently reported causes of pain include manipulation of the cervix with the tenaculum, uterine distension, application of hysteroscopic instruments, and performance of hysteroscopic procedures such as endometrial sampling. Some factors further enhance the degree of pain experienced, such as nulliparity, post-menopausal status, cervical stenosis and high anxiety level. On such occasions, the procedure has to be re-arranged in the operation theatre under regional or general anesthesia. Therefore, improvement in pain management can reduce patients' health care experience, patients' anesthetic and procedural risks, decrease healthcare costs, and reduce inconvenience to patients.

The major pain relief modalities include pharmacological and non-pharmacological techniques. The common analgesic agents used are non-steroid anti-inflammatory drugs (NSAID) and opioids; use of which is limited by their contraindications and side effects, such as deranged renal function and nausea. Non-pharmacological options are therefore a safer alternative. Some studies show that music and virtual reality are effective pain control for out-patient hysteroscopy. To date, there was only one published randomized controlled trial regarding the effectiveness of virtual reality in pain management. The study was limited by small sample size and conducted in only one center.

This randomized controlled trial aims at evaluating the effectiveness of non-pharmacological interventions (virtual reality and music therapy) in pain management during hysteroscopy. It can hopefully provide more clinical data to explore the role of non-pharmacological techniques in outpatient hysteroscopy pain control, hence help improve our participants' experience in outpatient hysteroscopy.

Objective:

This aim of the randomized controlled trial is to evaluate the effectiveness of non-pharmacological interventions (virtual reality or music therapy) in pain management based on the Numerical Pain Rating Scale (0-10) at different time-point of the hysteroscopy.

Study protocol:

Participants who meet the inclusion criteria will be introduced to the study by a female research assistant on the day of consultation.

During the consultation, participants' demographic data, obstetric and gynecological histories are obtained by the attending gynecologist using standardized datasheet. Consent for the hysteroscopy will be obtained according to the current practice. There will not be any routine prescriptions of analgesics to participants in the current standard practice.

Participants who are eligible for the study will be explained about the study, and written consent will be obtained by the attending gynecologist. Participants will be asked to rate their anticipated overall pain of outpatient hysteroscopy using a Numerical Pain Rating Scale (0-10), with 0 being no pain and 10 being the most severe pain.

Participants will be randomly assigned using sealed envelopes to 3 groups: (1) virtual reality group, or (2) music group, or (3) control group (current standard practice with no pain relief during the outpatient hysteroscopy procedure). Randomization will be carried out by using block randomization method with 1:1:1 ratio in block size of 6 and stratified by menopausal status (premenopausal or post-menopausal) and vaginal delivery (no vaginal delivery or history of vaginal delivery). Due to the nature of the intervention, both the investigators and the participants are not blinded to the allocation.

All participants will get ready for the diagnostic hysteroscopy on the gynecological examination bed as usual.

Participants assigned to the Visual reality group will be given the virtual reality device (a headset) with immersive video content for use during the hysteroscopy. Designated moving objects with sound will be broadcasted on the screen to the participant in this group. Participants in the music group will be given a headphone playing either classical light music or 'POP' songs according to their option during the hysteroscopy. Both groups of participants can adjust the volume of the sound or music according to her comfort. Disposable hygiene masks will be used as an underlay below the headset or headphone. Participants are allowed to stop the video or music, remove the headset or headphone at their own discretion or in the event of side effects. While participants in the control group will not be given any device.

The attending gynecologist will then perform the diagnostic hysteroscopy according to the standard procedures. Generally, a 30-degree hysteroscopy with normal saline as distending medium will be inserted through the cervical os into the uterine cavity under vision. No cervical dilation is required unless the hysteroscope is failed to enter the uterine cavity. The uterine cavity will be explored systematically. The procedure usually lasts for less than 10 minutes. If there is any endometrial pathology, the attending gynecologist will perform a targeted biopsy using the biopsy forceps. If there is no gross endometrial pathology, the diagnostic hysteroscope will be withdrawn and followed by endometrial aspirate to obtain endometrium for microscopic diagnosis if clinically indicated.

If there is/are small endometrial polyps (less than 1 cm), the attending gynecologist may perform excision of the polyp (polypectomy) by a hysteroscopic scissors, followed by retrieval of the polyp with biopsy forceps. Whether to proceed with polypectomy depends on the assessment of the operative feasibility by the attending gynecologist. If there is an indication to insert or remove an intrauterine contraceptive device, the procedure will be performed by the attending gynecologist. The indicated surgical procedure will not be affected by this trial.

If there is large endometrial polyp or submucosal fibroid not feasible for outpatient removal, participant will be arranged a hysteroscopic surgery under anesthesia later. The usual practice on management of these participants will not be affected by this trial.

Participants will be asked by the attending nurse to rate their pain score from 0 to 10 at different time-point of hysteroscopy; with 0 being no pain and 10 the most severe pain.

The duration of the whole diagnostic hysteroscopy is defined by the time of insertion of hysteroscope into the cervical os till withdrawal of the hysteroscope which will be recorded.

After the outpatient hysteroscopy, participants will be asked if they have experienced any side effects during the procedure. Besides, they will be asked to rate their satisfaction of the outpatient hysteroscopy, the communication with the attending gynecologist and staff during the hysteroscopy, their acceptance towards outpatient hysteroscopy in the future if indicated, and their recommendations to friends who may be indicated for outpatient hysteroscopy. Finally, they will be asked to rate the pain score 30 minutes after their procedure. Follow-up appointment or further treatment will be given to participant, if indicated, and not be driven by this trial.

ELIGIBILITY:
Inclusion Criteria:

* Participants scheduled for outpatient hysteroscopy in Prince of Wales Hospital
* Participants who are willing to give written consent to participate in the study

Exclusion Criteria:

* Participants who have hearing or visual deficits
* Participants who cannot understand written Chinese
* Participants refuse to participate in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2022-09-21 (Actual); Primary Completion 2023-07-05 (Actual); Study Completion 2023-07-05 (Actual)

PRIMARY OUTCOMES:
The change of the pain score of virtual reality therapy compared to control group (no intervention) in outpatient hysteroscopy. | Passage of hysteroscope through cervical internal os and during the assessment of uterine cavity of each participant. The study will be up to 1.5 years.
  The change of the pain score of virtual reality therapy at different time-point during outpatient hysteroscopy, compared to control group (no intervention).
  Pain score from 0 to 10, with 0 being no pain and 10 the most severe pain.
The change of the pain score of music therapy compared to control group (no intervention) in outpatient hysteroscopy. | Passage of hysteroscope through cervical internal os and during the assessment of uterine cavity of each participant. The study will be up to 1.5 years.
  The change of the pain score of music therapy at different time-point during outpatient hysteroscopy, compared to control group (no intervention).
  Pain score from 0 to 10, with 0 being no pain and 10 the most severe pain.

CONTACTS AND LOCATIONS:
Overall Officials: KA MAN YiP, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No